CLINICAL TRIAL: NCT00442923
Title: Scientific Component IV: Pharmacotherapy to Prevent Methamphetamine Relapse
Brief Title: "The Evaluation of Stimulant Withdrawal"
Acronym: MARC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was withdrawn for lack of progress. No subjects were recruited.
Sponsor: Aaron J. Janowsky (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Aaron J. Janowsky, Director, Methamphetamine Abuse Research Center, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1P50DA018165 (NIH); 1P50DA018165 (NIH)
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Anxiety; Relapse; Substance Addiction
Keywords: Methamphetamine; Coreg; Withdrawal; anxiety; Substance Addiction
MeSH Terms: conditions — Anxiety Disorders; Recurrence; Substance-Related Disorders | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CTRL (Placebo Comparator)
  Interventions: Drug: Coreg
- TREAT (Experimental)
  Interventions: Drug: Coreg

INTERVENTIONS:
Drug: Coreg

SUMMARY:
The purpose of this research study is to determine whether Carvedilol, an FDA approved beta blocker, when administered for an 8-week period to veterans currently undergoing treatment for methamphetamine dependence (1) improves their ability to stay in treatment longer, (2)eases the aversive symptoms that accompany stimulant withdrawal, and (3) increases the time they remain abstinent from methamphetamine.

ELIGIBILITY:
Inclusion Criteria:

* Must have entered treatment into the outpatient Clinical Addiction Rehabilitation Section (CARS) through the US Portland Veterans Affairs Medical Center
* Must meet the clinical definition for methamphetamine dependence
* Self-reported methamphetamine use within 10 days of entering the study
* Must be able to understand and sign the consent form

Exclusion Criteria:

* Dependent on any other drug except nicotine, caffeine, marijuana and alcohol
* Pregnant or nursing mothers
* Psychosis
* Dementia
* Any serious medical condition that could be aggravated by the study protocol (Allergic reaction, Hypotension, Asthma, Bronchospastic conditions, Angina, Bronchitis, Emphysema, Bradycardia, Heart or blood vessel disease, Diabetes mellitus, Low blood sugar, Kidney disease, Liver disease or Overactive thyroid)
* History of withdrawal seizures or delirium tremors
* Use of MAO inhibitors within the last two weeks
* Considerable hepatocellular injury, including cirrhosis of the liver or liver function test levels higher than 2 times normal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07-01 (Estimated); Primary Completion 2010-06-30 (Estimated); Study Completion 2011-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Berger, M.D., Principal Investigator — OHSU/ US VA
Locations (1):
- US Veterans Hospital, Portland, Oregon, United States